CLINICAL TRIAL: NCT07241260
Title: Boosting Brain and Mood: Exploring the Impact of Hydrate Heroes on Mental Health and Brain Activity
Brief Title: Hydrate Heroes for Improving Brain Function & Mood
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY008933; FHT-25-11 (Other Grant/Funding Number: Florida High-Tech Corridor)
Record Dates: First submitted 2025-07-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Hydration Status
Keywords: hydration; electroencephalography; EEG; brain activity; electrolytes; mental health; supplement; depression; anxiety
MeSH Terms: conditions — Psychological Well-Being; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hydrate Heroes A (Active Comparator): 6 packets / day
  Interventions: Dietary Supplement: Hydrate Heroes (6 packets)
- Hydrate Heroes B (Active Comparator): 3 packets / day
  Interventions: Dietary Supplement: Hydrate Heroes (3 packets)
- Control (No Intervention)

INTERVENTIONS:
Dietary Supplement: Hydrate Heroes (6 packets) — Participants that are randomized to the active comparator groups will receive 6 packets of Hydrate Heroes to use daily.
  Arms: Hydrate Heroes A
Dietary Supplement: Hydrate Heroes (3 packets) — Participants that are randomized to the active comparator groups will receive 3 packets of Hydrate Heroes to use daily.
  Arms: Hydrate Heroes B

SUMMARY:
The primary goal of this 12-week randomized controlled study is to evaluate whether daily use of Hydrate Heroes results in measurable improvements in brain activity, mental health, and performance on cognitive tasks. By analyzing brainwave data, physical response metrics, and patient-reported outcomes, the study will demonstrate whether the supplement produces meaningful effects on mental and neurological health.

DETAILED DESCRIPTION:
The study will utilize electrophysiological measurements of the brain and body.

EEG recordings will be captured using the Emotiv FLEX 2.0 wireless headset, which measures brainwave activity across 32 electrode sites using a standard 10-10 system. EEG data will be collected at 256 Hz and analyzed using EEGLAB software to assess spectral power and topographic changes over time. The protocol includes 20 minutes of EEG testing per session, with specific tasks designed to elicit measurable cognitive responses.

Participants will wear an Empatica Embrace wristband during testing to collect physiological data including motion, stress indicators, and heart rate variability.

Participants will complete a series of validated tests on an iPad while wearing the EEG headset and wrist device. Tasks include:

* Grandfather Passage (speech task)
* Card Matching (memory and attention)
* Boston Naming Test (language)
* Finger Tapping (motor speed)
* Trail Making Test (executive function)
* Dual-Task Performance (cognitive load)

Over 500 digital data features will be captured per session using a system that combines inputs from device sensors (e.g., gyroscope, camera, microphone) with user interactions (e.g., tapping, speech, app use).

Participants will complete standardized questionnaires, including PROMIS-29+2 and IPAQ-SF, to assess aspects such as emotional well-being, physical activity, fatigue, and pain. The PROMIS-29+2 is aA collection of short forms or computer adaptive tests containing a fixed number of items from seven PROMIS domains (Depression, Anxiety, Physical Function, Pain Interference, Fatigue, Sleep Disturbance, and Ability to Participate in Social Roles and Activities) The PROMIS-29+2 is used to calculate a preference score. Preference-based scores provide an overall summary of health-related quality of life on a common metric. Preference-based scores summarize multiple domains on a metric ranging from 0 (as bad as dead) to 1 (perfect or ideal health). Scores can be used in comparisons across groups and for cost-utility analyses. The profile includes all items in the PROMIS-29 Profile v2.1 plus two Cognitive Function Abilities items. T-scores from the measure can be used to calculate a preference-based score.

International Physical Activity Questionnaire (IPAQ) short form is an 8-item questionnaire that encompasses time spent walking, in moderate and vigorous physical activity. The short form is feasible to administer and shows similar reliability and validity results in comparison to the long form. Test-rest reliability indicates good stability and high reliability (α <.80). Scoring provides a categorization of low, moderate, or high intensity of physical activity. Ideally, this will be performed pre- and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years at time of consent.
* Fluent in English (able to read, write, speak, and understand English).
* Generally healthy, without chronic medical conditions (see Exclusion 10.3).
* Willing and able to attend three in-person study visits over an approximate 12-week period (enrollment, ~6 weeks, ~12 weeks).
* Willing to consume assigned Hydrate Heroes packets as directed (6 sticks/day, 3 sticks/day, or no supplement for control).
* Willing to log daily water intake and number of Hydrate Heroes packets consumed in the study's online tracking system.
* Capable of providing informed consent.

Exclusion Criteria:

* Neurological or Psychiatric Conditions
* History of epilepsy, recurrent seizures, severe head injury, or other significant neurological disorders.
* Current diagnosis of major psychiatric disorders (e.g., schizophrenia, bipolar disorder, severe major depressive disorder).

  · Cardiovascular or Renal Conditions
* Chronic kidney disease, congestive heart failure, or any condition requiring medically supervised fluid restriction.
* Documented electrolyte imbalance (e.g., hyponatremia, hypokalemia) within the past 6 months.
* Medication and Supplement Conflicts
* Use of medications known to alter EEG readings (e.g., benzodiazepines, antiepileptics, antipsychotics).
* Use of high-dose diuretics or other drugs that substantially affect hydration status.
* Concurrent use of any supplements containing one or more key ingredients of Hydrate Heroes - adaptogenic mushroom blends, magnesium, potassium, zinc, vitamin D₃, vitamin C (including Amla), electrolytes, or elderberry - that cannot be safely discontinued for the 12-week study duration.
* Reproductive Status
* Pregnant or currently breastfeeding.
* Compliance Risk
* Inability or unwillingness to reliably follow the hydration/supplement protocol or complete daily logging.
* Inability to attend scheduled visits or follow instructions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Electroencephalography - Frequencies | 12 weeks
  Measurement of brain electrical activity.
  Measures will include power band analysis (e.g., delta, theta, alpha, beta, gamma) summed over activities and comparisons made between groups (i.e. ratios).
Electroencephalography - ERP Amplitude | 12 weeks
  Measurement of brain electrical activity.
  Event-related potentials will be determined from events that occur during the activities. Differences in P300 amplitude will be determined (uV).
Electroencephalograpy - ERP Latency | 12 weeks
  Measurement of brain electrical activity.
  Event-related potentials will be determined from events that occur during the activities. Differences of P300 latency will be determined between groups (msec).

SECONDARY OUTCOMES:
Patient Reported Outcomes Measurement Information System (PROMIS)-29 + 2 | 12 weeks
  This single form patient reported outcome provides insight to pain, depression, anxiety, sleep, and physical function.
  Score will be reported as a t-score. The average t-score is 50. Deviation from 50 demonstrates magnitude of difference in either positive or negative direction.
International Physical Activity Questionnaire - Short Form (IPAQ-SF) | 12 weeks
  Patient reported outcome of physical activity over a 7-day period. The scores provide both a categorical output of 'Inactive', 'Slightly Active', and 'Active' and a continuous variable of metabolic equivalent (MET).

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Florida, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Michael J, John T, Templeton M. Towards a Comprehensive Mobile-Based Neurocognitive Digital Health Assessment System (NDHAS) Towards a Comprehensive Mobile-Based Neurocognitive Digital Health Assessment System (NDHAS) Templeton. J M. Published online 2022.
- [Background] Templeton JM, Poellabauer C, Schneider S. Design of a neurocognitive digital health system (NDHS) for neurodegenerative diseases. In: Proceedings of the 2021 Workshop on Future of Digital Biomarkers. ACM; 2021:26-33.
- [Background] Pion-Tonachini L, Kreutz-Delgado K, Makeig S. ICLabel: An automated electroencephalographic independent component classifier, dataset, and website. Neuroimage. 2019 Sep;198:181-197. doi: 10.1016/j.neuroimage.2019.05.026. Epub 2019 May 16. PMID 31103785
- [Background] Palmer JA, Kreutz-Delgado K, Makeig S. AMICA: An Adaptive Mixture of Independent Component Analyzers with Shared Components.
- [Background] Walters KF, Shukla R, Kumar V, Schueren S, Yadav H, Schilaty ND, Jain S. Resting-State EEG Power Spectral Density Analysis Between Healthy and Cognitively Impaired Subjects. Brain Sci. 2025 Feb 10;15(2):173. doi: 10.3390/brainsci15020173. PMID 40002506
- [Background] Delorme A, Makeig S. EEGLAB: an open source toolbox for analysis of single-trial EEG dynamics including independent component analysis. J Neurosci Methods. 2004 Mar 15;134(1):9-21. doi: 10.1016/j.jneumeth.2003.10.009. PMID 15102499
- See also: Hydrate Heroes - Main Webpage — https://hydrateheroes.com/?srsltid=AfmBOoqif6eNp5F4joMcwfmuMf625c_6VWruFip_v48r1zYNhu7BnXXX